CLINICAL TRIAL: NCT02741609
Title: A Multicenter Study to Evaluate a Borrelia Diagnostic Test in Subjects With Early Stage or Late Stage Lyme Disease
Acronym: ALSIBDT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor lack of funding
Sponsor: Advanced Laboratory Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IR-12
Record Dates: First submitted 2016-04-06; First posted 2016-04-18 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Lyme Disease
Keywords: Borrelia; spirochetes; culture; immunostaining
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Early/Late Stage Lyme disease (Experimental): Have early Lyme disease based on the following criteria: Signs, symptoms and clinical history consistent with early stage Lyme disease. Subjects must have a physician-diagnosed erythema migrans (EM) rash and should have systemic symptoms indicative of disseminated infection. Symptoms may include fever, headache, fatigue, myalgias, arthralgias, and stiff neck. Paired acute and convalescent titers will be drawn (first draw at time of initial visit and second draw 4 weeks later). Have late Lyme disease based on the following criteria: Signs, symptoms and clinical history consistent with late stage Lyme disease, including but not limited to disseminated rash, arthritis, meningitis, facial palsy, or carditis. Qualified subjects will be administered the Borrelia Diagnostic Test.
  Interventions: Device: Borrelia Diagnostic Test

INTERVENTIONS:
Device: Borrelia Diagnostic Test — The ALSI BDT is a high-yield in vitro cultivation method for Borrelia burgdorferi from venous whole blood samples.

SUMMARY:
This study will evaluate Advanced Laboratory Services Borrelia diagnostic test by culturing Borrelia spirochetes from human serum in subjects with early or late Lyme disease.

This is an 8 month study. Subjects entering the study will have two blood samples collected one month apart if they have early Lyme disease and one blood sample collected if they have late Lyme disease. Subjects who sign an IRB-approved consent form and meet the inclusion and exclusion criteria will be entered into the study. Subjects will be assigned a subject number upon entry and this number will be retained throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to the conduct of any study-related procedures.
2. Male or female subjects who are at least 18 years of age.
3. Subjects are suspected to have early Lyme disease based on the following criteria: Signs, symptoms and clinical history consistent with early-stage Lyme disease. Subjects must have a medical practitioner-diagnosed erythema migrans (EM) rash and should have systemic symptoms indicative of disseminated infection. Symptoms may include fever, headache, fatigue, myalgias, arthralgias, and stiff neck. Paired acute and convalescent titers will be drawn (first draw at time of initial visit and second draw 4 weeks later) or,
4. Subjects are suspected to have late Lyme disease based on the following criteria: Signs, symptoms and clinical history consistent with late stage Lyme disease, including but not limited to disseminated rash, arthritis, meningitis, facial palsy, or carditis.
5. Subjects must be willing and have the ability to safely have the required quantity of blood drawn for the study at the discretion of the investigator.
6. Subjects must have blood samples freshly collected (no supplemental frozen samples) and the samples must reach ALSI's laboratory on a weekday and within 24 hours of being drawn.

   ---

Exclusion Criteria:

1. Early Lyme disease: Subjects without an EM rash or do not have symptoms recognized as being associated with Lyme disease.
2. Exposure to antibiotics of any type during the 6 weeks prior to the initial blood sample collection.
3. Immune deficiency significant enough to render serological tests less reliable.
4. The subject is unwilling or unable to safely have the required quantity of blood drawn for this study.
5. Subjects who are not able to understand all of the requirements of the study or unable to give informed consent and/or comply with all aspects of the evaluation.
6. Subjects that have any other condition or situation which, in the opinion of the investigator, would make the subject unsuitable for enrollment or could interfere with the subject participating in and completing the study.
7. Subjects that have undergone testing for Lyme disease within the past year.
8. Subjects that have a prior diagnosis of Lyme disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the Advanced Laboratory Services, Inc. (ALSI) Borrelia Diagnostic Test (BDT) culture, for positive and negative predictive value, as compared to conventional microbiological methods. | Baseline to 16 weeks

SECONDARY OUTCOMES:
Diagnostic accuracy of ALSI culture for early-onset presentation of Lyme disease, as measured by positive and negative predictive value. | Baseline to 16 weeks
Diagnostic accuracy of ALSI culture for late-onset presentation of Lyme disease, as measured by positive and negative predictive value. | Baseline to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jasbir Arora, PhD, Principal Investigator — Advanced Laboratory Services
Locations (16):
- United States (16):
  - Delaware Integrative Medicine, Georgetown, Delaware
  - Penobscot Bay Medical Center, Rockport, Maine
  - Infectious Disease/The Research Institute, Springfield, Massachusetts
  - Birch Tree Healing Arts, Saint Paul, Minnesota
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Dr. Steven Bock, MD, Rhinebeck, New York
  - Dr. Marina Makous, Exton, Pennsylvania
  - Detweiler Family Medicine & Associates, PC, Lansdale, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Cumberland Valley Parochial Medical Clinic, Shippensburg, Pennsylvania
  - Lyme Center of New England, Cumberland, Rhode Island
  - The Miriam Hospital of Infectious Diseases, Providence, Rhode Island
  - Virginia Center for Health & Wellness, Aldie, Virginia
  - Rockbridge Traditional Medicine, Lexington, Virginia
  - Andrs Wellness Consulting, Petersburg, Virginia
  - Cardinal Internal Medicine, Woodbridge, Virginia

IPD SHARING:
Plan to Share IPD: No